CLINICAL TRIAL: NCT06334887
Title: A RCT of a Mobile App (esTOCma) to Improve Mental Health Literacy, Stigmatizing Attitudes Related to OCD, and Confidence in Dealing With Students With OCD in Teachers
Brief Title: esTOCma, an App Used by Teachers: an RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Principal Investigator, Gemma García-Soriano, PhD, associate professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PID2021-124409OB-I00_O3
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; adolescence; mobile app; mental health literacy; teachers
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: A parallel randomized controlled trial (RCT) with two arms: experimental group (use of esTOCma) and control group (untreated) will be carried out.
  As participants enroll in the study, those that meet the inclusion criteria will be randomized into experimental or control group and into contamination or aggressive vignette (see Outcome Measures). Everyone will complete the baseline measures (T1). Then, those assigned to experimental group will use the app esTOCma until they finish it (they will be given a 10-days deadline), whereas control group will do nothing for 10 days. After that, all the participants will complete again the assessment instruments (T2).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use of esTOCma (Experimental): Experimental group will use esTOCma until they finish it (within a preestablished 10-days period).
  Interventions: Device: Use of esTOCma
- Control group (No Intervention): Control group will do nothing for 10 days.

INTERVENTIONS:
Device: Use of esTOCma — Participants of the experimental group will use the esTOCma mobile app until completion, within a set period of 10 days.
  EsTOCma is a a serious game with 10 missions where users have to free 10 characters who have been imprisoned by a monster called esTOCma, which metaphorically represents the stigma in OCD. With each mission, users will gain knowledge about OCD and free an imprisoned character until the tenth mission, when they will defeat the monster. This game has three modules: (1) Psychoeducation (missions 1-5), where general information about OCD, OCD treatments and where to seek help is provided; (2) Indirect Contact (missions 6 and 7), which consists of a series of audio-visual recordings in which OCD patients report their symptoms and the impact the disorder has had on their lives; and finally, (3) Cognitive Restructuring (missions 8-10), where common dysfunctional beliefs about OCD and OCD treatment are challenged.
  Arms: Use of esTOCma

SUMMARY:
The aim of the present study is to assess the efficacy of a mobile application called esTOCma in promoting mental health literacy, reducing stigmatizing attitudes related to the Obsessive-Compulsive Disorder (OCD) and improving teachers' confidence in dealing with students that might have OCD. A parallel, randomized controlled trial with two conditions (experimental and control group) will be carried out in a sample of teachers that work in primary and secondary education. Pre-post changes will be assessed. Experimental group will use the app until they finish it (within a set period of 10 days), whereas control group will do nothing for 10 days. Primarily, it is expected that after the use of the app, participants will show an improvement in OCD-related literacy, stigmatizing attitudes, desired social distance and their comfort, confidence and perceived ability in teaching and handling students with OCD. Secondarily, the investigators hypothesize that experimental group might show a reduction in obsessive-compulsive symptoms.

DETAILED DESCRIPTION:
Adolescence is a critical stage that is associated with a high vulnerability to developing obsessive-compulsive disorder (OCD). Schools are part of the natural developmental context of adolescents, and teachers are involved in their education and personal development. In this sense, teachers play an essential role in the early detection and referral of students with possible obsessional symptoms and will also have to deal with the management of this symptomatology in the classroom. Moreover, teachers often have low knowledge of mental health problems and lack strategies for handling mental symptomatology in the classroom.

esTOCma is a mobile health (mHealth) application that has been developed to promote mental health literacy and reduce stigmatizing attitudes associated with OCD. Previous studies have shown that it is a tool with great potential in terms of intervention on stigma and OCD literacy in the general population. Thus, it could be of great interest to use this app in the field of education, and especially in non-university education since adolescents, a highly vulnerable collective to the development of OCD, spend much of their time in the classroom, and often seek help from school staff.

ELIGIBILITY:
Inclusion Criteria:

* Being a practising teacher in non-university education.
* Working in the education field as a guidance counsellor, language teacher or therapeutic pedagogue.

Exclusion Criteria:

* Working in a field other than those mentioned above.
* Having less than 18 years old.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in general OCD literacy | Through app completion (an estimation of 10 days).
  Score change in the knowledge and the attitudes towards obsessive-compulsive disorder measured by the OCD Knowledge Stigma Assessment Scale (OKSAS). It is a self-report ad hoc questionnaire with 24 items and a response scale ranging from 1 "Completely disagree" to 5 "Completely agree". The total score is the sum of the items and higher score indicate more knowledge about the disorder.
Change in stigmatizing attitudes related to OCD | Through app completion (an estimation of 10 days).
  Score change in stigma will be measured, in association with a vignette, by two questionnaires:
  1. Attribution Questionnaire (AQ-9; Corrigan et al., 2015; Spanish version: Muñoz et al., 2015) is a self-report measure for social stigma. It has a Likert scale ranging from 1 = "Not at all" to 9 = "Very much". Investigators will not use the items corresponding to Coercion, Pity and Avoidance. The higher the score (total and per item), the higher the stigma.
  2. OCD Stigma Measure (OSM; Ponzini et al., 2023) is a self-report measure composed by 16 items that assess OCD-related stereotypes. 11 items will be used in this study. A total score (sum of all the items) is interpreted.
  There will be two vignettes that will be randomly assigned. Both portray a student with OCD but one focuses on the contamination content, and the other on the aggression content.
Change in desired social distance | Through app completion (an estimation of 10 days).
  Score change in desired social distance will be measured by Reported and Intended Behaviour Scale (RIBS; Evans-Lacko et al., 2011; Spanish version: Sayols-Villanueva et al., 2015). It is a self-report measure with 8 items and it inquires about reported and intended behaviour among four different contexts: (1) living with, (2) working with, (3) living nearby and (4) continuing a relationship with someone with a mental health problem. Investigators will use the 4 items corresponding to intended behaviour subscale. Likert scale from 1 "Agree strongly" to 5 " Disagree strongly" and an additional "Don't know" response option. The total score is calculated by adding together the response values, and "Don't know" is coded as a neutral value (i.e. 3).
  This questionnaire will be used in association with a vignette.
Change in percieved confidence when addressing students with OCD | Through app completion (an estimation of 10 days).
  Score change in confidence when addressing students with OCD will be measured using items adapted and translated from previous studies (Jorm et al., 2010; Kutcher et al., 2016; Whitley & Gooderham, 2016). Three dimensions are evaluated separately:
  Confidence in interacting, composed of three items with a Likert scale ranging from 1 "Completely disagree" to 5 "Completely agree". The total score will be obtained by summing the item responses.
  Confidence in helping, assessed with a single item ("To what extent do you feel capable of helping a student like N?") rated on a 5-point scale ranging from 1 "Slightly/Not at all confident" to 5 "Extremely/Very confident".
  Academic confidence, measured with two items rated on a 4-point Likert scale ranging from 1 ("Not at all capable/ Lower academic level") to 4 ("Very capable/Highest academic level"). A total score will be computed by summing both items.

SECONDARY OUTCOMES:
Change in obsessive-compulsive symptoms | Through app completion (an estimation of 10 days).
  Score change in OCD symptoms will be measured by Obsessive-Compulsive Inventory - Revised. The reduced 4-item version (OCI-4; Abramovich et al., 2021) that assesses four dimensions of OCD (washing, checking, ordering, obsessing) will be used. It has a 5-point Likert scale ranging from 0 "Not at all" to 4 "Very much". The items will be added.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma García-Soriano, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia/ Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Share all IPD that underlie results in a publication.
Time Frame: It will be available for 3 months after the publication of the study.
Access Criteria: Data will be available in a repository website: Zenodo.
URL: https://zenodo.org/

REFERENCES:
- [Background] Chaves A, Arnaez S, Castilla D, Roncero M, Garcia-Soriano G. Enhancing mental health literacy in obsessive-compulsive disorder and reducing stigma via smartphone: A randomized controlled trial protocol. Internet Interv. 2022 Jul 13;29:100560. doi: 10.1016/j.invent.2022.100560. eCollection 2022 Sep. PMID 35874968
- [Background] Garcia-Soriano G, Arnaez S, Chaves A, Del Valle G, Roncero M, Moritz S. Can an app increase health literacy and reduce the stigma associated with obsessive-compulsive disorder? A crossover randomized controlled trial. J Affect Disord. 2024 Apr 1;350:636-647. doi: 10.1016/j.jad.2024.01.168. Epub 2024 Jan 20. PMID 38253133
- See also: Blog about the app esTOCma — http://estocma.es